CLINICAL TRIAL: NCT02116179
Title: DVD-based HIV/HCV Intervention for Drug-Involved Latino Criminal Justice Clients
Brief Title: DVD-based HIV/HCV Prevention Intervention for Drug-Involved Latino Criminal Justice Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R34DA031063 (NIH); 5R34DA031063 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Hepatitis C
Keywords: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Hepatitis C; Hispanic; Criminal Justice
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DVD Intervention (Experimental): DVD Intervention presented at one 90 minute group session
  Interventions: Behavioral: DVD Intervention
- Wait list Control Group (No Intervention): Group will get no intervention until after 90 day follow up

INTERVENTIONS:
Behavioral: DVD Intervention — Participants will be randomly assigned, with a baseline and 3 month follow up assessments
  Arms: DVD Intervention

SUMMARY:
The purpose of the study are the following: 1) Pilot test and conduct baseline and 3 month follow up assessments to evaluate the preliminary efficacy of the DVD-based HIV/HCV intervention by randomly assigning 210 Latino corrections-involved, outpatient abuse treatment clients to either the experimental intervention or to a wait list control group; and 2) to evaluate both participant and interventionist acceptability of this novel DVD-based intervention.

They study hypothesis are the following:

1. participants in the intervention condition will report greater reductions in sexual risk behaviors (e.g., unprotected sexual contact) from baseline to 3 month follow-up compared to the control group;
2. participants will report greater reductions in drug risk behaviors (e.g., sharing injection equipment, drug use during sex) from baseline to 3 month follow-up compared to the control group;
3. participants who report more HIV prevention information, motivation, and behavioral skills will report fewer sexual risk behaviors.

DETAILED DESCRIPTION:
The specific aims for Stage1b are: (1) to pilot test and evaluate the effectiveness of the DVD-based HIV intervention by recruiting 210 Latino offenders mandated to substance abuse treatment; and (2) to evaluate both participant and interventionist acceptability of this novel DVD intervention. Participants will be recruited from a local community agency that provides outpatient substance abuse treatment services for court-mandated individuals. Eligible participants will be self-identified Latino/Hispanic, between the ages of 18 and 49, heterosexual, and all participants will be involved with the criminal justice system. Participants will be randomized into either an intervention or a wait-list control condition. The intervention consists of one DVD-based group session facilitated by an interventionist. Sexual risk, drug use, mental health, and background information will be assessed at baseline, and again at 3 months after the intervention session. At the end of the intervention session, each participant will complete an acceptability questionnaire, and the interventionist will complete a checklist to assess treatment fidelity. It is hypothesized that both sexual risk and drug use behaviors will decrease between baseline and follow-up for the intervention group compared to the control group. The project is innovative because it will develop a DVD-based, culturally-appropriate and language specific, HIV/Hepatitis C virus prevention intervention for Latino offenders. The proposed research is significant, because it is expected to produce a brief HIV/Hepatitis C virus intervention that can be implemented within the criminal justice system and targets a high risk group.

It is hypothesized that participants in the intervention condition will report significant reductions in sexual risk behaviors (e.g., unprotected sexual contact) and drug risk behaviors (e.g. sharing injection equipment, drug use while having sex) from baseline to 3 - month follow-up when compared to control group. The main analysis here is to compare the proportion (or mean) of primary outcomes for those measured at 3-month (post-intervention) to those measured at baseline (pre-intervention) between the intervention and control group. The null is that there will be no differences, and alternative hypotheses would be that the intervention group will report more of a reduction in risk behaviors than control group. These hypotheses can be tested by either repeated-measures ANCOVA or regression with the robust cluster estimator obtained after controlling for intervention condition.

ELIGIBILITY:
Inclusion Criteria:

* must be between 18 - 49 years of age
* self-identify as Hispanic or Latino
* be involved in the criminal justice system
* report a history of drug use
* be in an outpatient substance abuse program
* self-identify as heterosexual

Exclusion Criteria:

* be HIV positive
* be cognitively impaired

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Sexual risk behaviors | 90 days

SECONDARY OUTCOMES:
Drug Use Behaviors | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gladys E Ibanez, PhD, Principal Investigator — Florida International University
Locations (1):
- University of Delaware Center for Drug and Alcohol Studies, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No